CLINICAL TRIAL: NCT02836626
Title: Fascial Scar Mobilization Techniques in Treating Chronic Caesarian Section Scar Pain: A Randomized Clinical Trial
Brief Title: Fascial Scar Mobilization Techniques in Treating Chronic Caesarian Section Scar Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rocky Mountain University of Health Professions (Other)
Collaborators: Franklin Pierce University (Other); Section on Women's Health American Physical Therapy Association (Unknown)
Responsible Party: Principal Investigator, Jennifer B. Wasserman, Assistant Professor, PhD candidate, Rocky Mountain University of Health Professions
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 160448-02
Record Dates: First submitted 2016-06-24; First posted 2016-07-19 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Cesarean Section; Cicatrix; Tissue Adhesions
MeSH Terms: conditions — Cicatrix; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Fascial Mobilization (Experimental)
  Interventions: Procedure: deep fascial mobilization
- Superficial Fascial Mobilization (Experimental)
  Interventions: Procedure: superficial fascial mobilization

INTERVENTIONS:
Procedure: deep fascial mobilization — Pelvic and abdominal myofascial release techniques as described by Barnes will be performed to facilitate independent mobility between tissue layers as needed following the direction of palpated fascial tension. Following this, direct scar mobilization techniques as described by Manheim will be done, applying a stretch in the direction of palpated restriction . This involves applying deep pressure whose force and direction is dictated by the tightness the therapist palpates and the subject reports. These are each held until a release is felt (defined as a sudden relaxation of tissue tension), usually 60-120 seconds. Total treatment time will last 25 minutes. Treatments will include all the above techniques but the therapist will tailor each treatment to address palpated restrictions. Subjects will be instructed to carry on their normal routines between sessions and will not be given any home interventions. Treatment sessions will total four to occur within a three week time period.
  Arms: Deep Fascial Mobilization
Procedure: superficial fascial mobilization — This group will undergo four 25-minute sessions of gentle superficial effleurage to the abdomen and posterior trunk followed by superficial skin rolling to the scar. Each treatment session will be terminated a) after 25 minutes or 2) when the patient asks to stop due to discomfort. Reasons for termination will be documented. Subjects will be instructed to carry on their normal routines between sessions and will not be given any home interventions. Treatment sessions will total four to occur within a three week time period.
  Arms: Superficial Fascial Mobilization

SUMMARY:
Over 1.37 million Caesarian sections (C-sections) are performed annually in the US . It is estimated that 12-20 % of those will result in chronic scar pain. This pain can lead to functional difficulties performing activities of daily living, pain with bowel movements, and pain with sexual activity . There is anecdotal evidence supporting the use of deep fascial scar mobilization techniques in reducing abdominal surgical scar pain, and yet almost no research has been published. The aims of this randomized clinical trial will be to determine if deep fascial scar mobilization techniques or superficial scar mobilization techniques will improve chronic pain and its resulting functional deficits, threshold pressure discomfort, pressure tolerance and mobility restrictions resulting from C-section surgery and to see if these interventions are more effective than no intervention. A positive result may result in an increase in the use of this intervention and thus the reduction of chronic scar pain for many women; it may provide justification for insurance reimbursement for this approach and it will also pave the way for further investigation into the use of these techniques with other types of painful scars including hysterectomy.

DETAILED DESCRIPTION:
Methods: Thirty six subjects will be recruited who have a history of C-section surgery more than three months before entering the study and who report chronic pain in or around the scar stemming from the surgery. Subjects will initially be tested twice four weeks apart, before beginning intervention. This will allow the establishment of a baseline and the subjects will all be part of a baseline control group. They will then be randomly assigned to one of two treatment groups. Group 1 will undergo four, 25 minute sessions of light massage to the trunk followed by superficial skin rolling of the C-section scar. Group 2 will undergo four, 25-minute treatment sessions consisting of multi-planar pelvic and abdominal myofascial mobilization techniques and direct scar mobilization techniques..

Outcomes: Outcome measures will include threshold pressure discomfort and pressure tolerance using a Pressure Algometer, Adheremeter measurements of scar mobility, the numeric pain rating scale (NPRS), the Oswestry Disability Index (ODI), Hip extension and shoulder flexion measured via goniometery, and the Global rating of Change scale. Follow up measures will be collected four weeks following the start of interventions and again at 12 weeks. In addition qualitative data will be collected from the subjects. The treating therapist will be blinded to the results of the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* well- healed abdominal scar over 3 months old that is resulting in chronic pain
* pain can be intermittent, at rest or with activity, and must have been present at least at a 3/10 at some point in the month prior to evaluation
* patient must report the presence of chronic pain.

Exclusion Criteria:

* history of cancer in pelvis or abdomen
* active infection / infectious disease in pelvis or abdomen
* pain medications on days of measurements
* skin irritation/inflammation at site of scar
* currently pregnant
* history of radiation to area
* Age <18
* no pain with pressure and mobility is symmetrical in all directions on initial examination.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Digital Pressure Algometer | Change from 0 weeks to 4 weeks to 8 weeks to 16 weeks
  6 points along the scar will be assessed. Pressure Pain threshold is the force (N) at which pressure turns to pain and Pressure Pain tolerance is the force (N) at which the pain becomes intolerable
Adheremeter | Change from 0 weeks to 4 weeks to 8 weeks to 16 weeks
  6 points along the scar will be assessed. Scar flexibility (mm) in each of 4 directions (superior, right, left, inferior) will be assessed at each point

SECONDARY OUTCOMES:
Global Rating of Change | Change from 4 weeks to 8 weeks to 16 weeks
  patient survey -7= very much worse; 0 = no change; +7= very much better
Goniometery hip extension and shoulder flexion | Change from 0 weeks to 4 weeks to 8 weeks to 16 weeks
Qualitative Assessment | change between 4 and 8 weeks during interventions
  subject comments as to response to interventions will be recorded for qualitative assessment
Numeric Pain Rating Scale | Change from 0 weeks to 4 weeks to 8 weeks to 16 weeks
  Subjects are asked to rate their pain in the past 48 hours and their current pain. Pain 0= no pain, 10= maximal pain
Oswestry Disability Index | Change from 0 weeks to 4 weeks to 8 weeks to 16 weeks
  Functional Index- patient survey

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Franklin Pierce University, Manchester, New Hampshire
  - ITR Physical Therapy, McLean, Virginia
  - Experience Momentum, Lynnwood, Washington